CLINICAL TRIAL: NCT00581997
Title: A Randomized, Double-blinded, Placebo Controlled, Multiple-dose, Multi-center Pilot Study, to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous Doses of QAX576 in Patients With Pulmonary Fibrosis Secondary to System Sclerosis
Brief Title: QAX576 in Patients With Pulmonary Fibrosis Secondary to Systemic Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Concerns about risk of bronchoscopy procedure in the selected patient population and frequency of SAEs observed to date.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAX576A2201
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2012-05

CONDITIONS: Pulmonary Fibrosis Secondary to Systemic Sclerosis
Keywords: Pulmonary fibrosis, systemic sclerosis
MeSH Terms: conditions — Pulmonary Fibrosis; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): QAX576
  Interventions: Drug: QAX576
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAX576
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will evaluate the safety, tolerability, and mechanism of action of multiple doses of QAX576 in patients with pulmonary fibrosis secondary to systemic sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18 and 65 years with a confirmed diagnosis of pulmonary fibrosis secondary to systemic sclerosis
* Both men and women must be willing to use two forms of contraception. Additional information regarding this requirement is available at screening

Exclusion Criteria:

* Certain medical conditions may exclude patients from participation.
* Should not have participated in another clinical study within 4 weeks of study start
* Smokers are not eligible for participation
* Blood loss of donation of 400 mL or more within 2 months of study start
* Pregnant women or women who are breast feeding
* Past medical history of clinically significant ECG abnormalities
* Connective tissue disorders other than systemic sclerosis.
* Active infection or history of systemic parasitic infection
* History of immunodeficiency diseases, including a positive HIV test result
* History of drug or alcohol abuse within 12 months of study start
* Any condition that may compromise patient safety

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
- Safety assessments including vital Signs, ECG's, Echocardiograms and blood draws. - The pharmacokinetics and pharmacodynamics of multiple doses of the drug will be assessed by blood draws at the 3 dosing visits. A blood sample will also be collected. | throughout the study

SECONDARY OUTCOMES:
- The effect of the drug on biomarkers of pulmonary fibrosis and systemic sclerosis. - Pulmonary function tests. - Disease specific measurements, active hand extension, oral aperture, MRSS. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Principal Investigator — Novartis Pharmaceuticals

REFERENCES:
- See also: Results for CQAX576A2201 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14398